CLINICAL TRIAL: NCT05062291
Title: Prospective, Multicenter, Observational Study to Evaluate the Merit WRAPSODY™ Endoprosthesis for Treatment of Stenosis or Occlusion Within the Dialysis Outflow Circuit of an Arteriovenous (AVF) Fistula or AV Graft (AVG) (The WRAP Registry)
Brief Title: Merit WRAPSODY™ Endoprosthesis for Treatment of Stenosis or Occlusion (WRAP)
Status: Active, not recruiting | Type: Observational
Sponsor: Merit Medical Systems, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CVO-P4-21-01
Record Dates: First submitted 2021-09-21; First posted 2021-09-30 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Venous Stenosis; Venous Occlusion
Keywords: Arteriovenous Fistula (AVF); Arteriovenous Graft (AVG); AV fistula; AV graft
MeSH Terms: conditions — Arteriovenous Fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Merit WRAPSODY Endovascular Stent Graft — Target Lesion Primary Patency (TLPP)

SUMMARY:
The WRAP Study aims to expand and understand the safety and efficacy data on the WRAPSODY Endoprosthesis System in a real-world population.

DETAILED DESCRIPTION:
Prospective, multicenter, observational study to evaluate the Merit WRAPSODY™ Endoprosthesis for treatment of stenosis or occlusion within the dialysis outflow circuit of an arteriovenous (AV) fistula or AV graft (The WRAP Registry)

ELIGIBILITY:
Inclusion Criteria:

1. Subject provides written informed consent for study participation.
2. Subject is male or female, with an age ≥ 18 years at date of enrollment.
3. Subject is willing to comply with site standard of care procedures and follow-up visit schedules over 24 months.
4. Subject is undergoing chronic hemodialysis with the hemodialysis access the intervention will be performed upon
5. The dialysis access is considered mature and has been used to deliver hemodialysis treatments for at least one session.
6. Subject has stenosis or occlusion within the dialysis outflow circuit of an arteriovenous (AV) fistula or AV graft and is treated with WRAPSODY Endoprosthesis System in accordance with device instructions for use.

Exclusion Criteria:

1. Subject has a planned surgical revision of access site.
2. Subject has a known or suspected infection of the hemodialysis access site, systemic infection and/or septicemia.
3. Subject has an uncorrectable coagulation disorder.
4. Known hypersensitivity to nickel titanium alloy.
5. Subject's hemodialysis access is anticipated to be abandoned within 6 months.
6. Subject is scheduled for kidney transplant or peritoneal dialysis within the next 6 months post-procedure.
7. Full expansion of a Percutaneous Transluminal Angioplasty (PTA) balloon cannot be achieved during predilatation.
8. Device would be placed in the Superior Vena Cava
9. Any inflow or outflow lesion that could jeopardize patency access long-term beyond the target treatment area.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The registry will include peripheral cases in both AV graft and AV fistula patients (including at the graft vein anastomosis of an AVG patient) and thoracic central patients in both AV graft and AV fistula patients.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-06-23 (Actual); Primary Completion 2026-04-15 (Estimated); Study Completion 2027-10-15 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with Target Lesion Primary Patency (TLPP) (Primary Effectiveness Endpoint) | 6 months
  Proportion of subjects with Target Lesion Primary Patency (TLPP) at 6 Months. TLPP is defined as freedom from clinically-driven target lesion revascularization (CD-TLR) or target lesion thrombosis measured through 6 months post-procedure, which is the time interval of uninterrupted patency after study procedure to the next intervention performed on the target lesion or uncorrectable target lesion occlusion.
Proportion of subjects without any localized or systemic safety events (Primary Safety Endpoint) | 30 days
  Proportion of subjects without any localized or systemic safety events through 30 days post-index procedure that affect the access or venous outflow circuit and resulted in reintervention, hospitalization, or death (not including stenosis or thrombosis).

SECONDARY OUTCOMES:
Proportion of subjects with Target Lesion Primary Patency | 12 and 24 months
  Proportion of subjects with Target Lesion Primary Patency
Proportion of subjects with Assisted Target Lesion Primary Patency (aTLPP) | 6, 12 and 24 months
  Proportion of subjects with Assisted Target Lesion Primary Patency (aTLPP)
Proportion of subjects with Access Circuit Primary Patency (ACPP) | 6, 12 and 24 months
  Proportion of subjects with Access Circuit Primary Patency (ACPP)
Rates of procedure- and device-related adverse events | Index procedure, 30 days, and months 6
  Rates of procedure- and device-related adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Dheeraj Rajan, MD, Principal Investigator — University of Toronto; Panagiotis Kitrou, Principal Investigator — University Hospital of Patras
Locations (35):
- Australia (5):
  - Monash Health, Clayton
  - Liverpool Hospital, Liverpool
  - Fiona Stanley Hospital, Murdoch
  - Sir Charles Gairdner Hospital, Nedlands
  - Princess Alexandra Hospital, Woolloongabba
- Brazil (14):
  - Hospital Felicio Rocho, Belo Horizonte
  - Afya Hospital, Brasília
  - Hospital Santa Lucia, Brasília
  - Hospital Vera Cruz, Campinas
  - Instituto Pro Renal, Curitiba
  - Complexo Hospitalar de Niterói, Niterói
  - Parana Medical Research Center, Paranã
  - Real Hospital Português de Beneficência em Pernambuco, Recife
  - Impar Servicos Hospitalares S/A - Hospital Sao Lucas, Rio de Janeiro
  - Rio de Janeiro State University, Rio de Janeiro
  - Hospital Da Bahia, Salvador
  - Centro Internacional de Pesquisa do Hospital Alemão Oswaldo Cruz, São Paulo
  - Hospital Santa Rita de Cassia, São Paulo
  - Instituto Dante Pazzanese de Cardiologia, São Paulo
- Germany (2):
  - Protestant Hospital Queen Elisabeth Herzberge, Berlin
  - University of Cologne, Cologne
- The General University Hospital of Patras, Rio, Greece
- Shaare Zedek Medical Center, Jerusalem, Israel
- Maastricht UMC+, Maastricht, Netherlands
- New Zealand (4):
  - Te Toka Tumai Auckland, Auckland
  - Te Whatu Ora Health NZ Waitemata, Auckland
  - Te Whatu Ora Health NZ Waitaha Canterbury, Christchurch
  - Te Whatu Ora Health New Zealand Waitemata, Hamilton
- CHUC - Centro Hospitalar e Universitário De Coimbra, Coimbra, Portugal
- United Kingdom (6):
  - Belfast City Hospital, Belfast Health and Social Care Trust, Belfast
  - Queen Elizabeth Hospital, University Hospital Birmingham, Birmingham
  - King's College Hospital, NHS Foundation Trust, London
  - Royal London Hospital, Barts Health NHS Trust, London
  - Churchill Hospital, Oxford University Hospitals NHS Foundation Trust, Oxford
  - Royal Berkshire NHS Foundation Trust, Reading

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rajan DK, Kitrou PM. Prospective, Multicenter, Observational Study to Evaluate a Cell-Impermeable Endoprosthesis for Treatment of Stenosis or Occlusion within the Dialysis Outflow Circuit of an Arteriovenous (AV) Fistula or AV Graft (The WRAP Registry). Cardiovasc Intervent Radiol. 2023 Sep;46(9):1285-1291. doi: 10.1007/s00270-023-03531-w. Epub 2023 Aug 17. PMID 37592020